CLINICAL TRIAL: NCT00651235
Title: A Randomized, Open-label, Active Control Trial to Evaluate the Effect of LOSARTAN Therapy on the Progression of Aortic Root Dilation in Patients With Marfan Syndrome
Brief Title: A Randomized, Open-label, LOSARTAN Therapy on the Progression of Aortic Root Dilation in Patients With Marfan Syndrome
Acronym: MFS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Mei -Hwan Wu, National Taiwan University Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 200610030M
Record Dates: First submitted 2008-03-03; First posted 2008-04-02 (Estimated); Last update posted 2010-06-09 (Estimated); Status verified 2010-06

CONDITIONS: Marfan Syndrome
MeSH Terms: conditions — Marfan Syndrome | interventions — Losartan; Atenolol; Propranolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- B (Experimental): In combination therapy,the maximal dose of Losartan is 100 mg/day for adult and 50 mg/day for children. 50 mg of Atenolol once daily, 20 mg of Propranolol twice daily for adult and 1 mg/Kg/day for children
  Interventions: Drug: Losartan and Atenolol or Propranolol
- A (Active Comparator): The maximal dose of Atenolol or Propranolol is 150 mg/day for adult and 2 mg/Kg/day for children.
  Interventions: Drug: Atenolol or Propranolol

INTERVENTIONS:
Drug: Losartan and Atenolol or Propranolol — 50 mg of Atenolol once daily, 20 mg of Propranolol twice daily for adult and 1 mg/Kg/day for children.
  Losartan is 100 mg/day for adult and 50 mg/day for children.
  Other Names: Cozaar and Tenormin or Inderal
  Arms: B
Drug: Atenolol or Propranolol — The maximal dose of Atenolol or Propranolol is 150 mg/day for adult and 2 mg/Kg/day for children.
  Other Names: Tenormin or Inderal
  Arms: A

SUMMARY:
To assess the efficacy of angiotensin II receptor blocker, Losartan, to prevent progressive dilation of aortic root in patients with Marfan syndrome.

DETAILED DESCRIPTION:
Marfan syndrome (MFS) is a multisystem connective tissue disorder of autosomal dominant inheritance1. The cardinal features are noted in the cardiovascular, ocular, and skeletal system. The most life-threatening complication of MFS is progressive aortic root dilation leading to aortic dissection or rupture. Losartan, an angiotensin II type I receptor (AT1) antagonist, is a drug already in clinical use for hypertension and type II diabetic nephropathy. A recent study showed that Losartan prevents aortic root dilation and lung problem in a mouse model of MFS. Therefore, the goals of this clinical trial are to examine the efficacy and safety of Losartan in patients with Marfan syndrome for aortic root dilation prevention.

ELIGIBILITY:
Inclusion criteria

* Marfan syndrome with recognized aortic root dilation
* Patients must be older than one year of age
* Beta-blocker treatment at least three months
* Must sign an informed consent form

Exclusion criteria

* Prior to aortic root surgery
* Aortic root dimension more than 5.5cm
* Aortic surgery within 6 months
* Diabetes mellitus or liver and renal dysfunction or asthma
* Pregnancy
* Intolerance to Losartan therapy

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2007-02; Primary Completion 2011-02 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Echocardiograms | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Mei-Hwan Wu, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Chiu HH, Wu MH, Wang JK, Lu CW, Chiu SN, Chen CA, Lin MT, Hu FC. Losartan added to beta-blockade therapy for aortic root dilation in Marfan syndrome: a randomized, open-label pilot study. Mayo Clin Proc. 2013 Mar;88(3):271-6. doi: 10.1016/j.mayocp.2012.11.005. Epub 2013 Jan 12. PMID 23321647